CLINICAL TRIAL: NCT03631238
Title: The Dual Impact of Homocysteine and Cholesterol on Cognitive Functions
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MWAmeen, Principle Investigator, Assiut University
Other Study IDs: Cholesterol and cognition
Record Dates: First submitted 2018-08-08; First posted 2018-08-15 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Hypercholesterolemia; Cognitive Dysfunction; Hyperhomocysteinemia
Keywords: Cholesterol; Dementia; Homocysteine; Cognitive dysfunctions
MeSH Terms: conditions — Hypercholesterolemia; Cognitive Dysfunction; Hyperhomocysteinemia; Dementia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Apparently normal participants: Participants are not complaining from any cognitive decline are subjected to cognitive and cholesterol and homocysteine levels assessment.
  Interventions: Diagnostic Test: Blood sampling for total cholesterol and homocysteine and cognitive assessment by psychometric tests.

INTERVENTIONS:
Diagnostic Test: Blood sampling for total cholesterol and homocysteine and cognitive assessment by psychometric tests. — all participant are subjected to cognitive assessment by psychometric tests by using the arabic version of Mini Mental State Exam (MMSE) and Memory Assessment Scale (MAS).
  Blood samples were collected in the morning using 10 mL yellow top (plain) Vacutainer tubes.
  Lipid profile (triglycerides, low-density lipoprotein (LDL), and high-density lipoprotein (HDL)) were measured by Assiut university labs using Cholesterol Kits and analyzed by COBAS Integra analyzer.
  Total cholesterol levels were calculated using the sum of the LDL and HDL plus one-fifth of triglyceride levels.
  Samples of serum homocysteine are collected, centrifuged to separate plasma within 30 minutes after venipuncture and stored in specialized container in the Department of Clinical Pathology at (-20◦C) temperature.
  Total homocysteine was measured by ELISA technique, Sinogen kits (Research Use Only) and Statfax-2100 microplate analyzer.

SUMMARY:
The study evaluates if the relationship between total serum cholesterol is dependent on the total serum homocysteine. Fasting blood samples will taken from participants and two batteries of cognitive scales will be used to asses any cognitive decline.

DETAILED DESCRIPTION:
The relationship between total serum cholesterol (TC) levels and cognition remains wily.

Some studies suggested that high TC level in old peoples is associated with a decreased risk of dementia.

Other studies have indicated that hypercholesterolemia may be a risk factor for cognitive decline and Alzheimer's disease (AD).

But a recent study published in 2014 by Cheng and colleagues, showed that, an inverse U-shaped relationship between total cholesterol level and cognitive score was found only in participants with normal homocysteine levels. Indicating that both low and high total serum cholesterol were associated with lower cognitive scores, ended to the relationship between cholesterol levels and cognitive function depends upon homocysteine levels, suggesting an interactive role between cholesterol and homocysteine on cognitive function in the elderly peoples.

The effect of high serum homocysteine (HHcy) levels on cognition was overwhelming regardless of the serum cholesterol levels but in peoples with normal homocysteine levels, both low and high cholesterol levels may be detrimental to cognitive health.

ELIGIBILITY:
Inclusion Criteria:

* Fifty hundred participants
* Participants are of both genders
* Aged 55 years old and over.

Exclusion Criteria:

* Patient with dementia.
* Renal and hepatic impairment.
* Parkinson's disease.
* Cerebrovascular stroke.
* Patient with chronic medical problems.
* Patients on statins.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included 41 participants, randomly selected from out-patient neurology and psychiatry clinics , Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
correlations between serum total cholesterol and homocysteine levels and cognitive functions | 1 hour
  Blood samples were collected after an overnight fast by using 10 mL plain tubes.
  Lipid profile was measured by using Cholesterol Kits and analyzed by COBAS Integra analyzer.
  Total cholesterol levels were measured using the sum of the LDL and HDL plus one-fifth of triglyceride levels.
  Samples of serum homocysteine (Hcy) are stored in specialized container at (-20◦C) temperature.
  Total Hcy was measured by ELISA technique, Sinogen kits and Statfax-2100 micro-plate analyzer.
  Cognitive functions were measured by using the Arabic version of: the 30 points Mini Mental State Exam (MMSE) and the Memory Assessment Scale (MAS) which consists of 12 subtests and the degree of 100 points.
  The mean of total MAS plus MMSE degrees is used (e.g., (100+30)/2=65 Points which is the maximum score).
  High, normal and low cholesterol level is compared to the mean of cognitive score only in participants with normal homocysteine levels (below 14 umol/l), higher levels of Hcy is excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Nageh F El Gamal, MD, Study Chair — Assiut University
Locations (1):
- Michael W Ameen, Asyut, Egypt

REFERENCES:
- [Background] de Champlain J, Wu R, Girouard H, Karas M, EL Midaoui A, Laplante MA, Wu L. Oxidative stress in hypertension. Clin Exp Hypertens. 2004 Oct-Nov;26(7-8):593-601. doi: 10.1081/ceh-200031904. PMID 15702613
- [Background] Burns JM, Honea RA, Vidoni ED, Hutfles LJ, Brooks WM, Swerdlow RH. Insulin is differentially related to cognitive decline and atrophy in Alzheimer's disease and aging. Biochim Biophys Acta. 2012 Mar;1822(3):333-9. doi: 10.1016/j.bbadis.2011.06.011. Epub 2011 Jul 1. PMID 21745566
- [Background] Cheng Y, Jin Y, Unverzagt FW, Su L, Yang L, Ma F, Hake AM, Kettler C, Chen C, Liu J, Bian J, Li P, Murrell JR, Hendrie HC, Gao S. The relationship between cholesterol and cognitive function is homocysteine-dependent. Clin Interv Aging. 2014 Oct 23;9:1823-9. doi: 10.2147/CIA.S64766. eCollection 2014. PMID 25364240
- [Background] Ansari R, Mahta A, Mallack E, Luo JJ. Hyperhomocysteinemia and neurologic disorders: a review. J Clin Neurol. 2014 Oct;10(4):281-8. doi: 10.3988/jcn.2014.10.4.281. Epub 2014 Oct 6. PMID 25324876